CLINICAL TRIAL: NCT05920954
Title: Urgent (<24 Hours) Versus Early (24 to 48 Hours) ERCP for Patients With Mild and Moderate Acute Cholangitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Urgent ERCP vs Early ERCP
Record Dates: First submitted 2023-05-23; First posted 2023-06-27 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2023-07

CONDITIONS: Acute Cholangitis
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Urgent ERCP (Experimental): Urgent ERCP (<24 Hours).
  Interventions: Procedure: ERCP
- Early ERCP (Experimental): Early ERCP(24 to 48 Hours).
  Interventions: Procedure: ERCP

INTERVENTIONS:
Procedure: ERCP — Repeat ERCP

SUMMARY:
Acute Cholangitis is an emergency associated with significant morbidity and mortality which require prompt recognition and treatment. The decompression of biliary tree along with antibiotics are mainstay of therapy. Randomized comparative studies showed that ERCP achieves biliary decompression with markedly less morbidity and mortality compared with surgery, regardless of clinical drainage. Percutaneous trans hepatic drainage (PTBD) can be alternative to endoscopic drainage in selected group especially advanced hilar strictures and patients who are unfit for endoscopic procedure.

Recent ASGE guidelines suggested the performance of ERCP within 48 hours for patients with acute cholangitis; however it is conditional recommendation with very low quality of evidence. Till date, no randomized trial has compared urgent ERCP versus early ERCP for acute cholangitis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met criteria for a definite diagnosis acute cholangitis.

Exclusion Criteria:

* Patients with severe acute cholangitis at admission.
* Age < 18 years.
* Pregnancy.
* Associated Acute Severe Pancreatitis.
* Patients with suspected high grade (Bismuth III/IV) biliary stricture in whom PTBD is considered as primary method of biliary drainage.
* Not giving consent.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-06-10 (Actual); Study Completion 2024-07-10 (Actual)

PRIMARY OUTCOMES:
ERCP performed within 24 hours of hospitalization versus ERCP performed between 24 to 48 hours of hospitalization | Two Years
  To perform a single-centre, randomized trial comparing the efficacy (the ability to produce a desired or intended result) of urgent versus early ERCP (Endoscopic retrograde cholangiopancreatography) for reducing the risk of 30 days of mortality.
ERCP performed within 24 hours of hospitalization versus ERCP performed between 24 to 48 hours of hospitalization | Two Years
  PRIMARY OUTCOME: 30 day mortality

SECONDARY OUTCOMES:
ERCP performed within 24 hours of hospitalization versus ERCP performed between 24 to 48 hours of hospitalization | Two Years
  1. Organ failure.
  2. In Hospital mortality.
  3. Hospital stay.
  4. Need for reintervention.
  5. Need for readmission.

CONTACTS AND LOCATIONS:
Locations (1):
- AIG Hospitals, Hyderabad, Telangana, India

IPD SHARING:
Plan to Share IPD: No